CLINICAL TRIAL: NCT05110989
Title: The CryoICE™ Cryoanalgesia Registry for Pain Management in Post-cardiothoracic Surgery Via Cryoablation of the Intercostal Nerves
Brief Title: A Multicenter Patient Registry on Outcomes From Cryoanalgesia of the Intercostal Nerves
Acronym: REDUCE
Status: Recruiting | Type: Observational
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: REDUCE2018
Record Dates: First submitted 2021-10-28; First posted 2021-11-08 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: AtriCure Cryo Nerve Block (cryoNB) Device Family — Use of Atricure Cryo Nerve Block Device Family to generate cryoanalgesia for the management of post operative pain.

SUMMARY:
This is a retrospective and prospective, multicenter, observational patient registry to record outcomes from patients undergoing cryoablation of the intercostal nerves (cryoanalgesia) for post-operative pain management.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose age is 12 years or above, and are able to give informed consent/assent specific to state and national law.
2. Patients have been scheduled by physician(s) to undergo or have undergone cryoablation of the intercostal nerves utilizing at least one AtriCure device or are similar patients treated without the use of cryoablation

Exclusion Criteria:

1. Patient is enrolled in a concurrent trial that may impact the treatment offered by the registry devices.
2. Patient with exclusion criteria required by local governance.
3. Women of childbearing potential who are, or plan to become, pregnant during the time of the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The REDUCE registry eligibility is open to sites and physicians performing cryo nerve block procedures as treatments for patients to generate croanalgesia as a post operative pain management method using the AtriCure Cryo Nerve Block (cryoNB) Device Family. Subjects must have been scheduled to undergo or have undergone the cryo nerve block procedure and must meet all eligibility criteria in order for their treatment and results to be considered for this registry.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-06-29 (Actual); Primary Completion 2035-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of cryo nerve block to generate cryoanalgesia as post operative pain management | From enrollment to 5 years after date of index procedure
  Collect pain score to assess the effect of cryoanalgesia effect with a follow up duration of up to 5 years.
Safety of cryo nerve block to generate cryoanalgesia as post operative pain management | From enrollment to 5 years after date of index procedure
  Collect adverse events occurred during and post operation to assess the safety of the cryo nerve block procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Curits Quinn, MD, Principal Investigator — Elliot Hospital
Locations (6):
- United States (6):
  - AdventHealth, Orlando, Florida
  - Henry Ford Health Rochester Hospital, Rochester, Michigan
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Elliot Hospital, Manchester, New Hampshire
  - The Christ Hospital, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No